CLINICAL TRIAL: NCT04333472
Title: Piclidenoson for Treatment of COVID-19 - A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Piclidenoson for Treatment of COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Collaborators: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-241COVID-19
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Coronavirus Infection
Keywords: Piclidenoson; CF101; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — CF101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Piclidenoson (Experimental): Piclidenoson 2 mg every 12 hours orally added to standard of care
  Interventions: Drug: Piclidenoson
- Placebo (Placebo Comparator): Placebo every 12 hours orally added to standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Piclidenoson — Piclidenoson 2 mg orally every 12 hours for up to 28 days
  Other Names: CF101
  Arms: Piclidenoson
Drug: Placebo — Placebo orally every 12 hours for up to 28 days
  Arms: Placebo

SUMMARY:
Patients with documented moderate COVID-19 infection will be randomized 1:1 to receive piclidenoson 2 mg Q12H orally with standard supportive care (SSC - intervention arm) or placebo orally with SSC (control arm) for up to 28 days.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, pilot trial of piclidenoson 2 mg Q12H added to SSC, compared to placebo plus SSC, in a population of hospitalized subjects with "Moderate" or "Severe" COVID-19 per U.S. National Institutes of Health (NIH) Coronavirus Disease 2019 (COVID-19) Treatment Guidelines (2020). Subjects will be randomized according to a 1:1 ratio to one of the trial arms, and treated for up to 28 days, at the discretion of the Investigator. Piclidenoson 2 mg and placebo are supplied as matching tablets for oral administration.

Following initial diagnosis of COVID-19, and after having provided informed consent, subjects will be randomized according to 1:1 ratio to one of the trial arms on Day 0. SSC will be implemented and documented for all subjects, and maintained throughout the treatment period.

Vital signs (temperature, blood pressure, pulse rate per minute, respiratory rate per minute, oxygen saturation (SpO2), and PaO2/FiO2) of subjects will be monitored twice daily according to SSC. Parameters of clinical, respiratory, and vital status will be collected daily. Viral shedding will be assessed on a regular basis. Samples for pharmacokinetic (PK) analysis will be collected on Day 4.

Efficacy of piclidenoson will be assessed by clinical, respiratory, and virologic parameters. Safety and tolerability of piclidenoson will be assessed by adverse event (AE) monitoring, vital signs assessment, electrocardiograms (ECGs), and clinical laboratory tests (complete blood count (CBC) and extended chemistry panel). Adverse events will be graded by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).

ELIGIBILITY:
Inclusion Criteria

1. Hospitalized subjects 18 to 85 years of age, inclusive
2. Able and willing to sign informed consent
3. Molecular (RT-PCR) diagnosis of SARS-CoV-2 infection
4. Moderate or Severe illness per NIH COVID-19 Treatment Guidelines:

   "Moderate" Illness:
   * Symptoms such as cough, fever, sore throat, malaise, myalgias, headache; and
   * Evidence of lower respiratory tract disease by clinical assessment and/or imaging; and
   * SpO2 >93% on room air at sea level

   "Severe" Illness, including any of the following:
   * Respiratory rate >30 breaths/minute; or
   * SpO2 ≤93% on room air at sea level; or
   * Ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300; or
   * Lung infiltrates >50% of pulmonary volume on imaging
5. Female subjects must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of investigational product
6. Female subjects of childbearing potential and male subjects with partners of childbearing potential must agree to use adequate methods of contraception during the study and through 90 days after the last dose of study medication. Female subjects of childbearing potential are all those except subjects who are surgically sterile, who have medically documented ovarian failure, or who are at least 1 year postmenopausal.

   1. For females: 2 of the following contraceptive methods, with at least 1 being a barrier method:

      * Hormonal contraceptives for at least 27 days before dosing
      * Intrauterine device (IUD) in place at least 27 days before dosing
      * Double-barrier methods (use of condom [male partner] with either diaphragm with spermicide or cervical cap with spermicide) from screening
      * Surgical sterilization of the partner (vasectomy at least 1 month before screening)
      * Female subjects must have a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of investigational product.
   2. For males: Surgical sterilization (vasectomy at least 1 month before screening) or double barrier methods.

Exclusion Criteria

1. 1. "Critical" Illness, per NIH COVID-19 Treatment Guidelines, including any of the following:

   * Respiratory failure; or
   * Septic shock; or
   * Multiple organ dysfunction
2. Subjects who require mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
3. Participation in another clinical trial concurrently
4. Concurrent treatment with immunomodulators or anti-rejection drugs
5. Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
6. History of any of the following diseases or conditions:

   * Advanced or decompensated liver disease (including presence or history of bleeding varices, ascites, encephalopathy, or hepato-renal syndrome)
   * Inability to swallow tablets, or gastrointestinal disease which could interfere with the absorption of piclidenoson
   * Any malignancy within 5 years before screening; exceptions are superficial dermatologic malignancies (e.g., squamous cell or basal cell skin cancer treated with curative intent)
   * Cardiomyopathy, significant ischemic cardiac or cerebrovascular disease (including history of angina, myocardial infarction, or interventional procedure for coronary artery disease), or cardiac rhythm disorder
   * QTcF interval on an average of triplicate ECGs >450 milliseconds (msec) for males or >470 msec for females (except when QT prolongation is associated with right or left bundle branch block, in which case enrollment is allowed)
   * Any condition which increases proarrhythmic risk, including hypokalemia, hypomagnesemia, congenital Long QT Syndrome
   * Ongoing or planned use of a concomitant medication that is on the CredibleMeds list of drugs known to cause Torsades de Pointes unless the subject can be screened and monitored under the guidelines proposed by Giudicessi (2020)
   * Pancreatitis
   * Severe or uncontrolled psychiatric disorder, e.g., depression, manic condition, psychosis, acute and/or chronic cognitive dysfunction, suicidal behavior, and relapse of substance abuse
   * Active seizure disorder defined by either an untreated seizure disorder or continued seizure activity within the preceding year despite treatment with anti-seizure medication
   * Bone marrow or solid organ transplantation
   * Any serious condition that, in the opinion of the investigator, would preclude evaluation of response or make it unlikely that the contemplated course of therapy and follow-up could be completed
7. Any of the following abnormal laboratory tests:

   * Platelet count <90,000 cells/mm3
   * Absolute neutrophil count (ANC) <1,500 cells/mm3
   * Estimated creatinine clearance (CrCl) <50 mL/min by Cockroft-Gault formulation
   * Bilirubin level ≥2.5 mg/dL unless due to Gilbert's syndrome
   * AST or ALT level ≥3X the upper limit of normal
   * Serum albumin level <3.0 g/dL
   * International normalized ratio (INR) ≥1.5 (except subjects maintained on anticoagulant medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects alive and free of respiratory failure | 29 days
  Proportion of subjects alive and free of respiratory failure (defined as need for non-invasive or invasive mechanical ventilation, high-flow oxygen, or extracorporeal membrane oxygenation) at Day 29
Proportion of subjects discharged home alive | 29 days
  Proportion of subjects alive and discharged to home without need for supplemental oxygen at Day 29
Treatment-emergent adverse events (AEs) | 29 days
  Proportion of patients experiencing AEs

SECONDARY OUTCOMES:
Clinical status | 29 days
  • Clinical status at Day 29 on NIAID 8-point ordinal scale (NIH 2020):
  1. Not hospitalized, no limitations
  2. Not hospitalized, with limitations
  3. Hospitalized, no active medical problems
  4. Hospitalized, not on oxygen
  5. Hospitalized, on oxygen
  6. Hospitalized, on high-flow oxygen or noninvasive mechanical ventilation
  7. Hospitalized, on mechanical ventilation or ECMO
  8. Death
Time to improvement | 29 days
  Time (days) to improvement of 2 points on 7-point ordinal clinical scale
Incidence of mechanical ventilation | 29 days
  Proportion of patients who require mechanical ventilation
Ventilator-free days | 29 days
  Ventilator-free days to Day 29
Incidence of Intensive Care Unit (ICU) admission | 29 days
  Proportion of patients who require ICU admission
Duration of ICU stay | 29 days
  Duration (days) of ICU stay
Time to hospital discharge | 29 days
  Time (days) to hospital discharge
Duration of need for supplemental oxygen | 29 days
  Duration (days) of need for supplemental oxygen
Time to virus negativity | 29 days
  Time (days) to virus negativity by RT-PCR, defined as absence of SARS CoV 2 on 2 consecutive days of sampling
SARS-CoV-2 viral load | 29 days
  SARS-CoV-2 viral load (number of copies) by quantitative RT-PCR
AEs leading to withdrawal | 29 days
  Proportion of patients experiencing AEs leading to early discontinuation of trial treatment
Treatment-emergent serious AEs (SAEs) | 29 days
  Proportion of patients experiencing SAEs
Treatment-emergent abnormalities in clinical laboratory parameters or electrocardiograms (ECGs) | 29 days
  Proportion of patients experiencing treatment-emergent changes in clinical laboratory parameters or ECGs
Incidence of meeting safety-related stopping rules | 29 days
  Proportion of patients who meet study safety-related stopping rules
Pharmacokinetics of piclidenoson in this patient population | 5 days
  Plasma concentrations over time of piclidenoson
Serum cytokine levels | 29 days
  Change from baseline in serum concentrations of cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Zivit Harpaz, Study Director — Can-Fite BioPharma Ltd
Locations (6):
- Bulgaria (2):
  - II Multiprofile Hospital for Active Treatment - Sofia EAD, Sofia
  - IV Multiprofile Hospital for Active Treatment - Sofia EAD, Sofia
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
- Romania (2):
  - Clinical Hospital for Infectious Diseases "St. Parascheva" Iasi, Iași
  - "Sfantul Ioan cel Nou" County Emergency Hospital Suceava, Suceava

IPD SHARING:
Plan to Share IPD: Yes
To be determined
Supporting Information: Study Protocol, CSR
Time Frame: January 2021, indefinitely
Access Criteria: To be determined

REFERENCES:
- [Background] Fishman P, Cohen S. The A3 adenosine receptor (A3AR): therapeutic target and predictive biological marker in rheumatoid arthritis. Clin Rheumatol. 2016 Sep;35(9):2359-62. doi: 10.1007/s10067-016-3202-4. Epub 2016 Feb 17. PMID 26886128
- [Background] Cohen S, Fishman P. Targeting the A3 adenosine receptor to treat cytokine release syndrome in cancer immunotherapy. Drug Des Devel Ther. 2019 Jan 30;13:491-497. doi: 10.2147/DDDT.S195294. eCollection 2019. PMID 30787591
- See also: Sponsor website — http://canfite.co.il